CLINICAL TRIAL: NCT00374868
Title: Phase 1/2 Study of Biweekly ALIMTA Plus Cisplatin in Patients With Locally, Advanced, Non-Resectable or Metastatic Urothelial Cancer
Brief Title: Pemetrexed Plus Cisplatin Bi-Weekly, in Patients With Urothelial Cancer (Metastatic, Locally Advanced or Non-Resectable)
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Eli Lilly and Company (Industry)
Responsible Party: Chief Medical Officer, Eli Lilly
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 8679; H3E-ES-S085 (Other: Eli Lilly and Company)
Record Dates: First submitted 2006-09-11; First posted 2006-09-12 (Estimated); Results first posted 2009-06-17 (Estimated); Last update posted 2010-11-04 (Estimated); Status verified 2010-10

CONDITIONS: Urologic Neoplasms
MeSH Terms: conditions — Urologic Neoplasms | interventions — Pemetrexed; Cisplatin

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Pemetrexed + Cisplatin (Experimental)
  Interventions: Drug: pemetrexed; Drug: cisplatin

INTERVENTIONS:
Drug: pemetrexed — Phase 1: 300 mg/m^2, intravenous (IV), days 1 and 15 every 28 days x 2 cycles (dose escalation: 300 mg/m^2, 400 mg/m^2, and 500 mg/m^2)
  Phase 2: phase 1 determined dose, intravenous (IV), days 1 and 15 every 28 days until disease progression, unacceptable toxicity or patient decision to discontinue or 6 cycles of therapy
  Other Names: LY231514; Alimta
Drug: cisplatin — Phase 1: 50 mg/m^2, intravenous (IV), days 1 and 15 every 28 days x 2 cycles
  Phase 2: 50 mg/m^2, intravenous (IV), days 1 and 15 every 28 days until disease progression, unacceptable toxicity or patient decision to discontinue or 6 cycles of therapy

SUMMARY:
To assess the anti-tumor activity, as measured by response rate to bi-weekly pemetrexed plus cisplatin, in chemo-naive patients with diagnosed metastatic or locally advanced (non-resectable) urothelial cancer.

ELIGIBILITY:
Inclusion Criteria:

* Histologically proven locally advanced disease or metastatic transitional cell carcinoma of the urothelium including bladder, urethra, ureter, and renal pelvis. Patients should not be suitable for surgery or radiation with curative intent. However patients whose pre-chemotherapy sites of disease are restricted to the primary or regional lymph node sites and who have a major response to chemotherapy will be evaluated for post-chemotherapy surgical resection of residual cancer if the tumor has become resectable at the end of chemotherapy.
* Measurable disease status, as defined in the Response Evaluation Criteria in Solid Tumors (RECIST) criteria (Therasse et al., 2000)
* One course of prior radiation therapy is allowed. Prior radiation must have been completed at least 4 weeks before enrolment into the study and the patients must have recovered from all toxic effects.

Exclusion Criteria:

* Have central nervous system (CNS) or leptomeningeal metastases (unless the patient has completed successful local therapy for CNS metastases and has been off corticosteroids for at least 4 weeks before starting study therapy). A screening computed tomography (CT) or magnetic resonance imaging (MRI) before enrollment in the absence of a clinical suspicion of brain metastases is not required.
* Inability to interrupt aspirin or other nonsteroidal anti-inflammatory agents 2 days before, the day of, and 2 days after the dose of pemetrexed plus cisplatin or cisplatin alone. If a patient is taking a nonsteroidal anti-inflammatory drug (NSAID) or salicylate with a long half-life (for example, naproxen, piroxicam, diflunisal) it should not be taken 5 days before the dose of pemetrexed (8-day period for long-acting agents such as piroxicam), the day of, and 2 days after the dose of pemetrexed plus cisplatin.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 59 (Actual)
Dates: Start 2006-08; Primary Completion 2008-04 (Actual); Study Completion 2008-04 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Call 1-877-CTLILLY (1-877-285-4559) Mon - Fri 9 AM - 5 PM Eastern Time (UTC/GMT - 5 hours, EST), Study Director — Eli Lilly and Company
Locations (5):
- Spain (5):
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Barcelona
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Madrid
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Pamplona
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Sabadell
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Santander

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: A total of 59 participants entered the trial (21 in Phase 1 and 38 in Phase 2). Phase 1 determined the dose for Phase 2 to be 400 mg/m^2. Phase 2 results are reported.
Groups:
- Pemetrexed + Cisplatin: Pemetrexed: phase 1 determined dose=400 mg/m2, intravenous (IV), days 1 and 15 every 28 days until disease progression, unacceptable toxicity or patient decision to discontinue or 6 cycles of therapy Cisplatin: 50 mg/m2, intravenous (IV), days 1 and 15 every 28 days until disease progression, unacceptable toxicity or patient decision to discontinue or 6 cycles of therapy
Period: Overall Study
Arm/Group | Pemetrexed + Cisplatin
Started | 38
Completed | 2
Not Completed | 36
Not completed — Adverse Event | 12
Not completed — Progressive Disease | 7
Not completed — Physician Decision | 13
Not completed — Lost to Follow-up | 1
Not completed — Death | 2
Not completed — Other - Not Specified | 1

BASELINE CHARACTERISTICS:
Arm/Group | Pemetrexed + Cisplatin
Number analyzed (Participants) | 38
Age Continuous [Mean (Standard Deviation); unit: years] | 67.1 (8.7)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 7
  Male | 31
Region of Enrollment [Number; unit: participants]
  Spain | 38
Eastern Cooperative Oncology Group (ECOG) Performance Status [Number; unit: participants] — Classifies patients according to their functional impairment. Scores range from 0 (Fully Active) to 5 (Death).
  participants
    0 - Fully Active | 21
    1 - Ambulatory, Restricted Strenuous Activity | 15
    2 - Ambulatory, No Work Activities | 2
Location of Primary Tumor [Number; unit: participants]
  Bladder | 32
  Ureter | 1
  Urethra | 1
  Renal Pelvis | 4
Height [Mean (Standard Deviation); unit: centimeters] | 166 (7.5)
Weight [Mean (Standard Deviation); unit: kilograms] | 77.4 (13.2)

OUTCOME MEASURES:

1. Primary Outcome: Best Overall Tumor Response
Description: Best response recorded from the start of treatment until disease progression/recurrence using Response Evaluation Criteria In Solid Tumors (RECIST) criteria that defines when participants improve ("respond"), stay the same ("stable"), or worsen ("progression") during treatment. Complete response (CR) = disappearance of all target lesions. Partial response (PR) = 30% decrease in the sum of the longest diameter of target lesions. Progressive disease (PD) = 20% increase in the sum of the longest diameter of target lesions. Stable disease (SD) = small changes that do not meet above criteria.
Time Frame: baseline to measured progressive disease (up to 620 days)
Measure: Number; unit: participants
Arm/Group | Pemetrexed + Cisplatin
Number analyzed (Participants) | 38
participants
  Complete Response | 2
  Partial Response | 13
  Stable Disease | 13
  Progressive Disease | 1
  Not Evaluated | 3
  Not Performed | 3
  Missing | 3

2. Secondary Outcome: Time to Response
Description: Defined as time from study enrollment to the first Complete Response or Partial Response (using RECIST criteria). Complete response (CR) = disappearance of all target lesions. Partial response (PR) = 30% decrease in the sum of the longest diameter of target lesions.
Time Frame: baseline to response (up to 620 days)
Population: 16 patients were censored.
Measure: Mean (Standard Error); unit: days
Arm/Group | Pemetrexed + Cisplatin
Number analyzed (Participants) | 38
days | 111.816 (6.480)

3. Secondary Outcome: Duration of Response
Description: The duration of a complete response (CR) or partial response (PR) was defined as the time from first objective status assessment of CR or PR to the first time of progression or death as a result of any cause. Complete response (CR) = disappearance of all target lesions. Partial response (PR) = 30% decrease in the sum of the longest diameter of target lesions.
Time Frame: time of response to progressive disease (up to 620 days)
Population: 10 patients were censored.
Measure: Mean (Standard Error); unit: days
Arm/Group | Pemetrexed + Cisplatin
Number analyzed (Participants) | 38
days | 184.100 (19.595)

4. Secondary Outcome: Duration of Stable Disease
Description: Defined as time from study enrollment to the first progression of disease, complete response, partial response, or death from any cause. Complete response (CR) = disappearance of all target lesions. Partial response (PR) = 30% decrease in the sum of the longest diameter of target lesions. Progressive disease (PD) = 20% increase in the sum of the longest diameter of target lesions. Stable disease (SD) = small changes that do not meet above criteria.
Time Frame: time of no response or progression (up to 620 days)
Population: 1 patient was censored.
Measure: Median (95% Confidence Interval); unit: days
Arm/Group | Pemetrexed + Cisplatin
Number analyzed (Participants) | 38
days | 80 [71 to 103]

5. Secondary Outcome: Time to Progressive Disease
Description: Defined as the time from study enrollment to the first date of disease progression. Time to disease progression was censored at the date of death if death was due to other cause. Progressive disease (PD) = 20% increase in the sum of the longest diameter of target lesions.
Time Frame: baseline to measured progressive disease (up to 620 days)
Population: 19 patients were censored
Measure: Mean (Standard Error); unit: days
Arm/Group | Pemetrexed + Cisplatin
Number analyzed (Participants) | 38
days | 260.182 (22.954)

6. Secondary Outcome: Time to Treatment Failure (TTF)
Description: Time from study enrollment to first observation of disease progression, death from any cause, or early discontinuation of treatment (including toxicity or if patient had stable disease after 4 cycles). TTF was censored at date of last follow-up visit for patients who did not discontinue early, who were still alive, and who had not progressed.
Time Frame: baseline to stopping treatment (up to 620 days)
Population: 1 patient was censored
Measure: Median (95% Confidence Interval); unit: days
Arm/Group | Pemetrexed + Cisplatin
Number analyzed (Participants) | 38
days | 133.5 [99 to 151]

7. Secondary Outcome: Progression-Free Survival
Description: Defined as the time from study enrollment until disease progression or death from any cause.
Time Frame: baseline to measured progressive disease (up to 620 days)
Population: 11 patients were censored
Measure: Median (95% Confidence Interval); unit: days
Arm/Group | Pemetrexed + Cisplatin
Number analyzed (Participants) | 38
days | 203 [137 to 285]

8. Secondary Outcome: Overall Survival
Description: Overall survival is the duration from enrollment to death. For patients who are alive, overall survival is censored at the last contact.
Time Frame: baseline to date of death from any cause (up to 620 days)
Population: 20 patients were censored.
Measure: Mean (Standard Error); unit: days
Arm/Group | Pemetrexed + Cisplatin
Number analyzed (Participants) | 38
days | 264.190 (15.130)

ADVERSE EVENTS:
Arm/Group | Pemetrexed + Cisplatin
Serious Adverse Events (participants affected / at risk) | 16
Other Adverse Events (participants affected / at risk) | 38
SERIOUS ADVERSE EVENTS; cells are participants affected / at risk (number of events):
Term (organ system) | Pemetrexed + Cisplatin
Anaemia (Blood and lymphatic system disorders) | 1/38 (3)
Febrile neutropenia (Blood and lymphatic system disorders) | 1/38 (1)
Leukopenia (Blood and lymphatic system disorders) | 3/38 (4)
Neutropenia (Blood and lymphatic system disorders) | 4/38 (5)
Thrombocytopenia (Blood and lymphatic system disorders) | 1/38 (1)
Cardio-respiratory arrest (Cardiac disorders) | 1/38 (1)
Abdominal pain (Gastrointestinal disorders) | 1/38 (1)
Diarrhoea (Gastrointestinal disorders) | 3/38 (3)
Dyspepsia (Gastrointestinal disorders) | 1/38 (1)
Nausea (Gastrointestinal disorders) | 2/38 (2)
Vomiting (Gastrointestinal disorders) | 3/38 (3)
Asthenia (General disorders) | 1/38 (1)
Pyrexia (General disorders) | 3/38 (3)
Pseudomonal sepsis (Infections and infestations) | 1/38 (1)
Urinary tract infection (Infections and infestations) | 3/38 (3)
Blood electrolytes abnormal (Investigations) | 1/38 (1)
Anorexia (Metabolism and nutrition disorders) | 1/38 (1)
Bone pain (Musculoskeletal and connective tissue disorders) | 1/38 (1)
Renal failure (Renal and urinary disorders) | 2/38 (2)
Renal impairment (Renal and urinary disorders) | 1/38 (1)
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 1/38 (2)
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 2/38 (2)
Deep vein thrombosis (Vascular disorders) | 4/38 (4)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected / at risk (number of events):
Term (organ system) | Pemetrexed + Cisplatin
Anaemia (Blood and lymphatic system disorders) | 8/38 (12)
Neutropenia (Blood and lymphatic system disorders) | 2/38 (3)
Thrombocytopenia (Blood and lymphatic system disorders) | 3/38 (7)
Tinnitus (Ear and labyrinth disorders) | 2/38 (2)
Conjunctivitis (Eye disorders) | 4/38 (4)
Abdominal discomfort (Gastrointestinal disorders) | 2/38 (3)
Abdominal pain (Gastrointestinal disorders) | 10/38 (10)
Abdominal pain lower (Gastrointestinal disorders) | 2/38 (2)
Abdominal pain upper (Gastrointestinal disorders) | 5/38 (5)
Constipation (Gastrointestinal disorders) | 10/38 (18)
Diarrhoea (Gastrointestinal disorders) | 18/38 (32)
Dry mouth (Gastrointestinal disorders) | 2/38 (2)
Dyspepsia (Gastrointestinal disorders) | 4/38 (4)
Nausea (Gastrointestinal disorders) | 20/38 (48)
Stomatitis (Gastrointestinal disorders) | 2/38 (4)
Tongue ulceration (Gastrointestinal disorders) | 2/38 (2)
Vomiting (Gastrointestinal disorders) | 20/38 (30)
Asthenia (General disorders) | 29/38 (82)
Chest pain (General disorders) | 2/38 (2)
Gait disturbance (General disorders) | 3/38 (3)
Mucosal inflammation (General disorders) | 14/38 (33)
Oedema (General disorders) | 4/38 (6)
Oedema peripheral (General disorders) | 6/38 (10)
Pyrexia (General disorders) | 3/38 (6)
Influenza (Infections and infestations) | 2/38 (2)
Nasopharyngitis (Infections and infestations) | 2/38 (2)
Urinary tract infection (Infections and infestations) | 2/38 (2)
Alanine aminotransferase increased (Investigations) | 2/38 (2)
Aspartate aminotransferase increased (Investigations) | 2/38 (2)
Gamma-glutamyltransferase increased (Investigations) | 2/38 (2)
Weight decreased (Investigations) | 2/38 (2)
Anorexia (Metabolism and nutrition disorders) | 19/38 (26)
Decreased appetite (Metabolism and nutrition disorders) | 4/38 (4)
Diabetes mellitus (Metabolism and nutrition disorders) | 2/38 (2)
Dyslipidaemia (Metabolism and nutrition disorders) | 2/38 (2)
Back pain (Musculoskeletal and connective tissue disorders) | 7/38 (8)
Limb discomfort (Musculoskeletal and connective tissue disorders) | 2/38 (2)
Musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 2/38 (2)
Pain in extremity (Musculoskeletal and connective tissue disorders) | 2/38 (2)
Dizziness (Nervous system disorders) | 3/38 (3)
Dysgeusia (Nervous system disorders) | 7/38 (12)
Headache (Nervous system disorders) | 3/38 (3)
Neuropathy (Nervous system disorders) | 2/38 (2)
Paraesthesia (Nervous system disorders) | 5/38 (10)
Tremor (Nervous system disorders) | 2/38 (2)
Depression (Psychiatric disorders) | 2/38 (2)
Insomnia (Psychiatric disorders) | 3/38 (3)
Dysuria (Renal and urinary disorders) | 3/38 (3)
Haematuria (Renal and urinary disorders) | 2/38 (2)
Cough (Respiratory, thoracic and mediastinal disorders) | 2/38 (3)
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 5/38 (6)
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 2/38 (2)
Hiccups (Respiratory, thoracic and mediastinal disorders) | 2/38 (2)
Erythema (Skin and subcutaneous tissue disorders) | 3/38 (4)
Pruritus (Skin and subcutaneous tissue disorders) | 2/38 (2)
Rash (Skin and subcutaneous tissue disorders) | 4/38 (4)
Deep vein thrombosis (Vascular disorders) | 2/38 (2)
Hypertension (Vascular disorders) | 5/38 (5)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of more than 60 days